CLINICAL TRIAL: NCT01610609
Title: Center for Advancing Equity in Clinical Preventive Services Project 2: Reducing Disparities in Primary Prevention of Cardiovascular Disease
Brief Title: Reducing Disparities in Primary Prevention of Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen Persell, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1P01HS021141-01-Project 2; 1P01HS021141-01 (NIH)
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Cardiovascular Diseases; Cholesterol, LDL
Keywords: Statin treatment; Cardiovascular disease; High cholesterol; Care management
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Population Health Management Intervention (Experimental): Participants randomized to this arm will receive the population health management intervention.
  Interventions: Behavioral: Population Health Management Intervention
- Usual Care Control Group (No Intervention): Participants randomized to this arm will receive usual care.

INTERVENTIONS:
Behavioral: Population Health Management Intervention — This intervention includes:
  * Care manager led patient education to promote increased patient awareness of personal cardiovascular disease (CVD) risk and
  * Care manager led patient outreach to facilitate the treatment of eligible and appropriate patients with statins for primary CVD prevention
  Arms: Population Health Management Intervention

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of disparities in years of life lost by race and low socioeconomic status. Statins have been shown to decrease the risk of cardiovascular events among individuals with high CVD risk. Yet, despite increased statin use and overall declining CVD rates, disparities in statin use and disparities in the control of high cholesterol by race, ethnicity, and socioeconomic status have persisted.

Objective: To improve the appropriate use of statins for primary cardiovascular disease prevention among high risk individuals at community health centers through a system of population health management that uses electronic health record (EHR) data to identify patients for targeted education and outreach.

Aim 1: Conduct a randomized controlled trial among individuals with 10-year risk for myocardial infarction or coronary death of 10% or higher to determine if the population health management intervention, compared to usual care, results in higher rates of documented statin treatment discussions within 6 months (primary process outcome), higher rates of statin prescribing within 6 months (secondary process outcome), and higher rates of significant low-density lipoprotein cholesterol (LDL-C) lowering defined as a follow up LDL-C ≥30 mg/dL lower than baseline (primary clinical outcome).

Aim 2: Interview patients who received the intervention to identify barriers to success

Aim 3: Assess the overall costs of the intervention and the costs per each patient who achieves significant LDL-C lowering compared to patient who received usual care.

ELIGIBILITY:
Inclusion Criteria:

* men >= 35 and women >= 45 years old
* LDL-C completed in the past 5 years
* Not currently prescribed lipid lowering medication
* >= 1 face to face visit to a study site in the 6 months prior to the start of the study or a visit during the enrollment period
* The 10-year risk of coronary death or myocardial infarction (based on Framingham Risk Score) is at least 10% and the LDL-C is above 100 mg/dL

Exclusion Criteria:

* Previously diagnosed with any of the following: coronary disease, peripheral arterial disease, carotid artery disease, abdominal aortic aneurysm, or diabetes mellitus
* Primary language is not English or Spanish

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Discussion between provider and patient about statin treatment | within 6 months of randomization
  We will use queries of the electronic health record to detect documentation of face-to-face or telephone discussions regarding statin treatment. Physician investigators will be blinded to study group status and categorize variable as YES if there is documentation of any of the following in the chart (1) prescription for a statin (2) recommendation for statin therapy (3) patient refusal of statin (4) discussion of the use of a drug to lower cholesterol.

SECONDARY OUTCOMES:
Statin prescription | within 6 months of randomization
  We will query the electronic health record to determine whether or not a statin was prescribed in the 6 months following randomization
Low-density lipoprotein cholesterol (LDL-C) | within 1 year of randomization
  We will query the electronic health record to determine whether there was a significant lowering of LDL-C defined as a follow up LDL-C >= 30 mg/DL lower than baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Persell, MD MPH, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - North Country Health Care, Flagstaff, Arizona
  - Near North Health Service Corporation, Chicago, Illinois
  - Heartland Health Outreach, Chicago, Illinois

REFERENCES:
- [Derived] Karmali KN, Lee JY, Brown T, Persell SD. Predictors of cholesterol treatment discussions and statin prescribing for primary cardiovascular disease prevention in community health centers. Prev Med. 2016 Jul;88:176-81. doi: 10.1016/j.ypmed.2016.04.011. Epub 2016 Apr 16. PMID 27090436
- [Derived] Persell SD, Brown T, Lee JY, Shah S, Henley E, Long T, Luther S, Lloyd-Jones DM, Jean-Jacques M, Kandula NR, Sanchez T, Baker DW. Individualized Risk Communication and Outreach for Primary Cardiovascular Disease Prevention in Community Health Centers: Randomized Trial. Circ Cardiovasc Qual Outcomes. 2015 Nov;8(6):560-6. doi: 10.1161/CIRCOUTCOMES.115.001723. Epub 2015 Nov 10. PMID 26555123